CLINICAL TRIAL: NCT04703127
Title: Effectiveness and Tolerability of the On-demand Use of Combined Dapoxetine With Tadalafil and Combined Dapoxetine With Lidocaine 5% Spray in Treatment of Patients With Lifelong Premature Ejaculation and Non-responding to Dapoxetine Alone.
Acronym: PE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Abu El-Hamd, Assistant Professor of Dermatology, Venereology and Andrology Department, Faculty of Medicine, Sohag University, Egypt., Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3/2020
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Premature Ejaculation
Keywords: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Tadalafil; Lidocaine

STUDY DESIGN:
Intervention Model Description: All patients will be equally divided into 2 groups (30 patients each). Group 1 was given on-demand 30 mg dapoxetine and 10 mg tadalafil 1 h before intercourse. Group 1 was given on-demand 30 mg dapoxetine 1 h before intercourse and apply lidocaine 5% spray on the glans penis 10 minutes the wash before intercourse.
Who Masked: Investigator
Masking Description: All patients will be equally divided into 2 groups (30 patients each).Group 1 was given on-demand 30 mg dapoxetine and 10 mg tadalafil 1 h before intercourse. Group 1 was given on-demand 30 mg dapoxetine 1 h before intercourse and apply lidocaine 5% spray on the glans penis 10 minutes the wash before intercourse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with lifelong premature ejaculation and non-responding to dapoxetine alone (Active Comparator): Group 1 was given on-demand 30 mg dapoxetine and 10 mg tadalafil 1 h before intercourse.
  Interventions: Drug: Tadalafil and Combined Dapoxietine
- Patients with Lifelong Premature Ejaculation and Non-responding to Dapoxetine Alone. (Active Comparator): Group 2 was given on-demand 30 mg dapoxetine 1 h before intercourse and apply lidocaine 5% spray on the glans penis 10 minutes the wash before intercourse.
  Interventions: Drug: Dapoxietine and Combined Lidocaine 5% Spray

INTERVENTIONS:
Drug: Tadalafil and Combined Dapoxietine — Group 1 was given on-demand 30 mg dapoxetine and 10 mg tadalafil 1 h before intercourse.
  Other Names: Tadalafil with Combined Dapoxietine
Drug: Dapoxietine and Combined Lidocaine 5% Spray — Group 2 was given on-demand 30 mg dapoxetine 1 h before intercourse and apply lidocaine 5% spray on the glans penis 10 minutes the wash before intercourse.
  Other Names: Dapoxietine With Lidocaine 5% Spray

SUMMARY:
Therefore, this study will aim to assess the effectiveness and tolerability of the on-demand use of combined dapoxetine with tadalafil and combined dapoxetine with lidocaine 5% spray in treatment of patients with lifelong premature ejaculation and non-responding to dapoxetine alone.

DETAILED DESCRIPTION:
This study will be carried out on 60 patients with lifelong premature ejaculation and non-responding to dapoxetine alone.

All patients will be equally divided into 2 groups (30 patients each). Group 1 was given on-demand 30 mg dapoxetine and 10 mg tadalafil 1 h before intercourse. Group 1 was given on-demand 30 mg dapoxetine 1 h before intercourse and apply lidocaine 5% spray on the glans penis 10 minutes the wash before intercourse.

ELIGIBILITY:
Inclusion Criteria:

* lifelong premature ejaculation and non-responding to dapoxetine alone.

Exclusion Criteria:

* diabetes mellitus,
* chronic prostatitis,
* Advanced renal or hepatic diseases
* neurological diseases
* C.N.S. medications

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male Patients with PE
Enrollment: 60 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Intravaginal ejaculatory latency time (IELT) | 0-8 weeks
Arabic Index of Premature Ejaculation (AIPE) | 0-8 week

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A El-Hamd, Principal Investigator — Dermatology, Venereology and Andrology, Faculty of Medicine, Sohag University
Locations (1):
- Mohammed Abu El-Hamd, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No